CLINICAL TRIAL: NCT03126123
Title: Assessment of the Predictive Value of the Acetic Acid Test in Surgery Condition for the Detection of Dysplastic Lesions in Patients With Anal Condylomatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0550
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Anal Condyloma
Keywords: Anal condylomatosis; surgery; acetic acid; dysplastic areas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acetic acid test (Other): Patients will receive surgical treatment for anal condylomatosis and acetic acid on the mucosa of the anal canal before the surgical procedure
  Interventions: Procedure: acetic acid test

INTERVENTIONS:
Procedure: acetic acid test — Patients will receive acetic acid on the mucosa of the anal canal before the surgical procedure

SUMMARY:
Anal condylomatosis is an anal canal mucosa pathology caused by HPV infection (Human Papilloma Virus). This condition is common, especially in immunodepressed patients.

These lesions are not accessible to topical medical treatment because of their location. They should be treated surgically because they may degenerate into squamous cell carcinoma.

In the operating room, lesions are identified by a complete proctologic examination, more or less supplemented by an acetic acid test. Acetic acid allows to detect mucous degeneration (dysplasia) in the form of intense bleaching. The interpretation of this test may nevertheless be difficult in case of local inflammation or scarring. These false positives may lead to unnecessary surgical gestures. The surgical procedure consists of a mucosectomy or destruction of the condylomatosis by electrocoagulation.

The acetic acid test is used at the discretion of the surgeon. However, there is little data on its performance or consensus on its use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* programmed surgery for anal condylomatosis in the visceral surgery department of the Hôpital de la Croix Rousse in Lyon
* patient in receipt of the social security scheme
* patient who did not oppose his participation in the study.

Exclusion Criteria:

* Pregnant women
* Patients protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of the acetic acid test in comparison with the anatomopathological analysis of the biopsies performed on the lesions revealed by acetic acid | the day of surgery
  Application of acetic acid just before surgery to identify suspect areas of dysplasia.
  Biopsies of suspicious areas bleached with acetic acid. The true positives (TP) will correspond to lesions bleached by acetic acid and showing dysplasia at biopsy. False positives (FP) will correspond to lesions bleached by acetic acid but not showing dysplasia at biopsy. The positive predictive value (PPV) will be the proportion of TP over the total number of bleached lesions. (PPV = TP / (TP + FP)). The PPV will be given with its 95% confidence interval (95%CI).

SECONDARY OUTCOMES:
Evaluation of the toxicity of the acetic acid test | the day of surgery
  Collection of adverse events associated with acetic acid use in peroperative time
Identify a patient subgroup in which the acetic acid test would be particularly discriminatory | up to 5 months before surgery
  Pre-surgery data collection on patient file at pre operative visit
post-surgery pain | up to 1 month post surgery
  self-assessed using a visual analog scale at 5; 12 hours post surgery;at Day 1; Day 2 ; Day 3; Day 7 ; Day 14; Day 21 post surgery; 1 month post-surgery
change in post-surgery incontinence | up to 5 months before surgery and 1 month post surgery
  evaluation with the Wexner score (anal incontinence score used internationally) before surgery (at pre operative visit) and 1 month post-surgery
Clinical recurrence of anal condylomatosis | 1 month post surgery
Duration of sick leave | 1 month post surgery
  number of days of sick leave
Number of unscheduled medical visits | 1 month post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Darnis, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital de la Croix Rousse, Lyon, France